CLINICAL TRIAL: NCT04866602
Title: A Randomised, Open Label 2-period Crossover Study to Evaluate the Relative Bioavailability of Atoguanil Compared to Malarone® in Healthy Adult Participants in the Fed State
Brief Title: Atoguanil BA Study
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Medicines for Malaria Venture (Other)
Collaborators: Richmond Pharmacology Limited (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: MMV_SMC_19_02
Record Dates: First submitted 2021-04-20; First posted 2021-04-30 (Actual); Last update posted 2022-05-05 (Actual); Status verified 2022-05

CONDITIONS: Bioavailability
Keywords: Pharmacokinetics; Bioavailability; Malaria prevention; Malaria
MeSH Terms: conditions — Malaria | interventions — atovaquone, proguanil drug combination

STUDY DESIGN:
Intervention Model Description: In Period 1, 16 participants will be enrolled and randomised to one of two treatments in a ratio of 1:1, and to the alternative treatment in Period 2, as described below:
  * Treatment 1: Single dose of Atoguanil . (Atovaquone 500 mg + Proguanil 348 mg administered as 4 tablets of 125 mg: 87 mg).
  * Treatment 2: Single dose of Malarone® . (Atovaquone 1000 mg + Proguanil HCl 400 mg administered as 4 tablets of 250 mg: 100 mg), Both doses are administered in the fed state and with 240mL of drinking water.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Atoguanil (Experimental): Atovaquone 500 mg + Proguanil 348 mg
  Interventions: Drug: Atoguanil
- Malarone® (Active Comparator): Atovaquone 1000 mg + Proguanil HCl 400 mg
  Interventions: Drug: Malarone

INTERVENTIONS:
Drug: Atoguanil — Atovaquone + Proguanil free base:125 mg: 87 mg, 4 tablets
  Other Names: Atovaquone + Proguanil
  Arms: Atoguanil
Drug: Malarone — Atovaquone + Proguanil HCl: 250 mg: 100 mg, 4 tablets
  Other Names: Atovaquone + Proguanil
  Arms: Malarone®

SUMMARY:
This trial aims to characterise the pharmacokinetic (PK) profile and estimate drug exposure from Atoguanil in comparison to Malarone®.

DETAILED DESCRIPTION:
After being informed about the study and potential risks, all adult participants giving written informed consent will be screened within 30 days prior to entering the trial on Day -1 to determine eligibility for study entry. The trial will establish whether the PK profile of both atovaquone (ATV), proguanil (PG) and cycloguanil (CG) from Atoguanil is similar to Malarone® and whether exposure of ATV from Atoguanil indicates that at least a 2-fold reduction in ATV dose compared with Malarone® is feasible (i.e. that the bioavailability of ATV in Atoguanil is approximately double that of ATV in Malarone®).

ELIGIBILITY:
Inclusion Criteria:

1. Healthy male or female (of childbearing and non-childbearing potential) aged 18 to 55 years, inclusive. Efforts will be made to ensure a reasonable gender balance.
2. Satisfactory medical assessment with no clinically significant or relevant abnormalities as determined by medical history, physical examination, vital signs and clinical laboratory evaluation (haematology, biochemistry, coagulation, and urinalysis) that is reasonably likely to interfere with the participant's participation in or ability to complete the trial as assessed by the Investigator.
3. Participant has a body weight of 50 to 80 kg and a body mass index (BMI) of 18.0-25.0 kg/m2, inclusive at screening.
4. All participants must comply with the contraception criteria in Section 5.5.
5. Participants must agree not to donate sperm or ova from the time of the first administration of trial medication until three months after the end of the systemic exposure of the trial drug (for this trial, this is until Day 22 of Period 2).
6. Participants are non-smokers (fewer than 100 lifetime cigarettes and zero cigarettes in the past 6 months).
7. Participants who are able to provide written, personally signed, and dated informed consent to participate in the trial, in accordance with the ICH Good Clinical Practice (GCP) Guideline E6 (R2) (2016) and applicable regulations, before completing any trial-related procedures.
8. Participants who are willing and able to comply with all scheduled visits, treatment plan, laboratory tests, restrictions, and other trial procedures. Participants must be willing to complete all meals, which may contain meat (in particular, the high fat, high calorie breakfast on dosing days).
9. Participants who are willing to comply with the latest site guidelines regarding COVID-19 safety precautions, measures and testing

Exclusion Criteria:

1. Female detected to be pregnant, breast feeding or who is likely to become pregnant during the trial.
2. Male participants with a female partner(s) who is (are) pregnant or lactating from the time of the administration of trial medication.
3. Evidence or history of clinically significant haematological, renal, endocrine, pulmonary, gastrointestinal, cardiovascular, hepatic, psychiatric, neurologic, or allergic disease (including drug or food allergies, anaphylaxis or other severe allergic reactions but excluding untreated, asymptomatic, seasonal allergies at the time of dosing).
4. Current or relevant history of physical or psychiatric illness (in particular, anxiety disorders) that may require treatment or make the participant unlikely to fully comply with the requirements or complete the trial, or any condition that presents undue risk from the investigational product or trial procedures.
5. Any surgical or medical condition possibly affecting drug absorption (e.g. cholecystectomy, gastrectomy, bowel disease, etc.), distribution, metabolism or excretion or any food intolerance.
6. Any other significant disease or disorder which, in the opinion of the Investigator, may either put the participant at risk because of the participation in the trial may influence the result of the trial, or the participant's ability to participate in the trial.
7. History of photosensitivity.
8. History or clinical evidence of substance and/or alcohol abuse within the 12 months before screening. Alcohol abuse is defined as regular weekly intake of more than 14 units for males and females (using alcohol tracker http://www.nhs.uk/Tools/Pages/NHSAlcoholtracker.aspx).
9. Treatment with an investigational drug within 90 days or 5 half-lives preceding the first dose of trial medication (or as determined by the local requirement, whichever is the longer).
10. Donation of blood or blood products (excluding plasma) within 90 days prior to trial medication administration.
11. Has used any medication listed on the Flockhart table (http://medicine.iupui.edu/clinpharm/ddis/main-table/) that is either a moderate or strong inhibitor or inducer of CYP450 within 30 days or 5 half-lives (whichever is longer) prior to the planned first day of dosing.
12. Additionally, participants must not have consumed other substances known to be potent inhibitors or inducers of CYP P450s . This includes food or drink products containing cranberry, pomegranate, star fruit, grapefruit, pomelos, exotic citrus fruits or Seville oranges (including marmalade and juices made from these fruits) in the two weeks before the planned first trial drug administration.
13. Has used any other prescription medication (excluding hormonal contraception, hormone replacement therapy) within 14 days or 10 half-lives (whichever is longer) prior to Day 1 of the dosing period that the Investigator judges is likely to interfere with the trial or pose an additional risk in participating.
14. Has used any over-the-counter medication (including multivitamin, herbal, or homeopathic preparations; excluding paracetamol - up to 4g paracetamol per day permitted) during the 7 days or 10 half-lives of the drug (whichever is longer) prior to Day 1 of the dosing period, that the Investigator judges is likely to interfere with the trial or pose an additional risk in participating.
15. Use of herbal supplements at least 30 days prior to the first dose of trial medication.
16. Known hypersensitivity reaction to atovaquone or proguanil.
17. Any clinically significant abnormal laboratory, vital signs or other safety findings as determined by medical history, physical examination or other evaluations conducted at screening or on admission.
18. The history or presence of any of the following cardiac conditions: known structural cardiac abnormalities; family history of long QT syndrome; cardiac syncope or recurrent, idiopathic syncope; exercise related clinically significant cardiac events.

1. Any clinically significant abnormalities in rhythm, conduction or morphology of resting ECG or clinically important abnormalities that may interfere with the interpretation of QTc interval changes. This includes participants with any of the following at screening:

1. Sinus node dysfunction.
2. Clinically significant PR (PQ) interval prolongation.
3. Intermittent second- or third-degree AV block.
4. Complete bundle branch block.
5. Sustained cardiac arrhythmia's including (but not limited to) atrial fibrillation or supraventricular tachycardia; any symptomatic arrhythmia with the exception of isolated extra systoles.
6. Abnormal T wave morphology which may impact on the QT/QTc assessment.
7. QT interval corrected using the Fridericia's formula (QTcF) > 450 ms (males and females).
8. Any other ECG abnormalities in the standard 12-lead ECG and 24-hour 12 lead Holter ECG or an equivalent assessment which in the opinion of the investigator will interfere with the ECG analysis. Participants with borderline abnormalities may be included if the deviations do not pose a safety risk, and if agreed between the appointed cardiologist and the investigator.

   Participants with borderline abnormalities may be included if the deviations do not pose a safety risk, and if agreed between the appointed Cardiologist and the PI.

   19. Confirmed positive results from urine drug screen (amphetamines, benzodiazepines, cocaine, cannabinoids, opiates, barbiturates, and methadone) or from the alcohol breath test at screening or on admission.

   20. A positive human immunodeficiency virus (HIV) I and II antibodies, hepatitis B surface antigen (HBsAg), anti-Hepatitis core antibody (anti HBc Ig G [and anti HBc IgM if IgG is positive]), or hepatitis C virus (HCV) antibody at screening.

   21. Participants have veins unsuitable for intravenous puncture or cannulation on either arm (e.g. veins that are difficult to locate access or puncture veins with a tendency to rupture during or after puncture).

   22. Participants with difficulty in swallowing multiple tablets at a time.

   23. Any conditions which in the opinion of the Investigator would make the participant unsuitable for enrolment or could interfere with the participants' participation in or completion of the trial.

   24. Participants who have received or are planning on receiving a COVID-19 vaccination as per section 6.3.1.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 16 (Actual)
Dates: Start 2021-11-17 (Actual); Primary Completion 2022-03-18 (Actual); Study Completion 2022-03-18 (Actual)

PRIMARY OUTCOMES:
Ratio of maximum observed plasma concentration (Cmax) of ATV, PG and CG from Atoguanil in comparison to Malarone. | ATV evaluation: Measured pre-dose -1 hours, then 1, 2, 2.5, 3, 3.5, 4, 4.5, 5, 6, 8, 10, 12, 16, 24, 48, 72, 168, 336, 504 hours post-dose. PG/CG evaluation: At pre-dose -1 then 1, 2, 2.5, 3, 3.5, 4, 4.5, 5, 6, 8, 10, 12, 16, 24, 48, 72 hours post-dose
  Blood samples are collected at indicated time points to measure the maximum observed plasma concentration (Cmax) for pharmacokinetic analysis of ATV, PG and CG. Pharmacokinetic parameters are determined using standard non-compartmental methods.
Ratio of the area under the plasma concentration-time curve from time zero to last detectable plasma concentration (AUC0-t) of ATV, PG and CG for Atoguanil compared to Malarone | ATV evaluation: Measured pre-dose -1 hours, then 1, 2, 2.5, 3, 3.5, 4, 4.5, 5, 6, 8, 10, 12, 16, 24, 48, 72, 168, 336, 504 hours post-dose. PG/CG evaluation: At pre-dose -1 then 1, 2, 2.5, 3, 3.5, 4, 4.5, 5, 6, 8, 10, 12, 16, 24, 48, 72 hours post-dose
  Blood samples are collected at indicated time points to measure the area under the plasma concentration-time curve from time zero to last detectable plasma concentration (AUC0-t) for pharmacokinetic analysis of ATV, PG and CG. Pharmacokinetic parameters are determined using standard non-compartmental methods
Ratio of area under the plasma concentration-time curve from time zero to 72 hours (AUC0-72h), of ATV, PG and CG for Atoguanil compared to Malarone. | Measured from 0 to 72 hours ATV/PG/CG evaluation: At pre-dose -1 and then 1, 2, 2.5, 3, 3.5, 4, 4.5, 5, 6, 8, 10, 12, 16, 24, 48, 72 hours post-dose
  Blood samples are collected at indicated time points to measure the area under the plasma concentration-time curve from time zero to 72 hours (AUC0-72h) for pharmacokinetic analysis of ATV, PG and CG. Pharmacokinetic parameters are determined using standard non-compartmental methods
Ratio of the area under the plasma concentration-time curve from time zero to 168 hours (AUC0-168h) [ATV only] for Atoguanil compared to Malarone | Measured from 0 to 168 hours (ATV) ATV evaluation: At pre-dose -1, and then 1, 2, 2.5, 3, 3.5, 4, 4.5, 5, 6, 8, 10, 12, 16, 24, 48, 72, 168 hours post-dose
  Blood samples are collected at indicated time points to measure the area under the plasma concentration-time curve from time zero to 168 hours (AUC0-168h) for pharmacokinetic analysis of ATV. Pharmacokinetic parameters are determined using standard non-compartmental methods.
Ratio of the area under the plasma concentration-time curve from time zero extrapolated to infinity (AUC0-inf), of ATV, PG and CG for Atoguanil compared to Malarone | ATV evaluation: Measured pre-dose -1 hours, then 1, 2, 2.5, 3, 3.5, 4, 4.5, 5, 6, 8, 10, 12, 16, 24, 48, 72, 168, 336, 504 hours post-dose. PG/CG evaluation: At pre-dose -1 then 1, 2, 2.5, 3, 3.5, 4, 4.5, 5, 6, 8, 10, 12, 16, 24, 48, 72 hours post-dose
  Blood samples are collected at indicated time points to measure the area under the plasma concentration-time curve from time zero extrapolated to infinity (AUC0-inf) for pharmacokinetic analysis of ATV, PG and CG. Pharmacokinetic parameters are determined using standard non-compartmental methods.

CONTACTS AND LOCATIONS:
Overall Officials: Ulrike Lorch, MD FRCA FFPM, Principal Investigator — Richmond Pharmacology Limited
Locations (1):
- Richmond Pharmacology Limited, London, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
De-Identified individual participant data for all primary and secondary outcome measures will be made available.
Supporting Information: Study Protocol
Time Frame: Data will be available within 6 months after study completion.
Access Criteria: Requestors will be required to sign a Data Access Agreement.

REFERENCES:
- [Derived] Kuemmerle A, Gossen D, Marx MW, Lorch U, Szramowska M, Kumar A, Singh D, Singh S, Ramachandruni H, Thankachen B, Kore S, Gaaloul ME, Borghini-Fuhrer I, Chalon S. A randomized, open-label two-period crossover pilot study to evaluate the relative bioavailability in the fed state of atovaquone-proguanil (Atoguanil) versus atovaquone-proguanil hydrochloride (Malarone(R)) in healthy adult participants. Naunyn Schmiedebergs Arch Pharmacol. 2024 Dec;397(12):9823-9832. doi: 10.1007/s00210-024-03245-x. Epub 2024 Jun 25. PMID 38918235